CLINICAL TRIAL: NCT01642433
Title: Prazosin as a Novel Treatment for Smoking Cessation
Brief Title: Prazosin for Smoking Cessation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Lung Association (Other)
Responsible Party: Principal Investigator, Christian Hendershot, Independent Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 071/2011
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar pills (Placebo Comparator)
  Interventions: Drug: Placebo
- Prazosin pills (Active Comparator)
  Interventions: Drug: Prazosin

INTERVENTIONS:
Drug: Placebo — Placebo capsules, 3x daily
  Arms: Sugar pills
Drug: Prazosin — Prazosin medication, 3x daily dosing, up to 15mg/day
  Arms: Prazosin pills

SUMMARY:
The most likely outcome of smoking cessation attempts is relapse, underscoring the need to advance novel treatments. Preclinical research shows that the noradrenergic system is critical for modulating drug-seeking behavior and recent findings indicate that the α1-adrenergic antagonist prazosin reduces nicotine self-administration and reinstatement. Presently, data on prazosin's effects on nicotine-related behaviour in humans is lacking. An efficient method for screening novel smoking cessation medications is to integrate human laboratory paradigms in the context of brief, randomized trials of smoking cessation that include smokers motivated to quit. This study aims to provide an initial test of prazosin for smoking cessation by implementing a brief, randomized trial that will include both human laboratory and clinical phenotypes. This approach will allow an efficient but sensitive method for medication screening that maximizes clinical validity.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 10 cigarettes per day for past year
* Baseline Fagerstrom Test for Nicotine Dependence (FTND) score of greater than or equal to four
* Willing to engage in two practice quit attempts
* Willingness to forgo other medication based treatments during the trial

Exclusion Criteria:

* Current illicit drug use
* Current treatment with psychiatric medications other than selective serotonin re-uptake inhibitors (SSRIs)
* Lifetime diagnosis of post-traumatic stress disorder (PTSD)
* Significant medical/neurological illness
* Baseline BP outside of normal range
* Current use of tobacco aids
* Current use of medications that could interact with prazosin
* Pregnancy or nursing

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Short-term smoking cessation | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Related Info — http://www.camh.net/research